CLINICAL TRIAL: NCT06543017
Title: Changes in Physiological Performance, Psychological State, and Sleep Quality of Athletes From Sichuan Province, China During the Pre Competition Weight Loss Stage
Brief Title: Pre Competition Weight Loss of Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chengdu Sport University (Other)
Responsible Party: Principal Investigator, Cheng Liang, Principal Investigator, Chengdu Sport University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SSC2024
Record Dates: First submitted 2024-08-01; First posted 2024-08-07 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Body Weight Changes
Keywords: wrestling; weight reduction; physiological performance; mental state; sleep quality
MeSH Terms: conditions — Body Weight Changes; Weight Loss; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: The participates of the study were 16 male freestyle wrestlers from Sichuan Province, China, preparing for the 2024 Chinese Wrestling Championships (4th to 12th May 2024). Based on their competition categories, they were to participate in five weight classes (57, 61, 65, 70, and 74 kg), with a total of 16 individuals (four in the 70 kg class, and three per other class). The study period was 38 days prior to the competition. Based on the training schedule and weight reduction characteristics, it was divided into a slow weight reduction phase (where athletes reduced weight slowly by adjusting their dietary structure and increasing the volume of aerobic exercise) and a rapid weight reduction phase (where athletes achieved rapid weight loss by further restricting water intake and adjusting their diet).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): A total of three tests were conducted on all participants, each time between 6:00 and 9:00 in the morning. The first test (first day of slow weight reduction, T1) was on 26th March, the second test (first day of rapid weight reduction, T2) was on 26th April, and the third test (the day before the competition, T3) was on 3rd May.
  Interventions: Other: Experimental group

INTERVENTIONS:
Other: Experimental group — This study included 16 male freestyle wrestlers from Sichuan Province, China. Participants were tested at three time points: the first day of slow weight reduction (T1), the first day of rapid weight reduction (T2), and the day before competition (T3), with measurements taken for physiological performance, mental state, and sleep quality.

SUMMARY:
The objective of this observational study is to assess the long-term impact of a combined slow and rapid weight reduction strategy on the physiological performance, mental state, and sleep quality of male freestyle wrestlers. The primary question it seeks to address is:

Does the combined weight reduction approach affect the physiological performance, mental state, and sleep quality of male freestyle wrestlers during the pre-competition period?

Participants will undergo tests at three stages of their weight reduction process (T1, T2, T3) over a period of 38 days prior to the competition, providing data on various physiological and psychological indicators.

DETAILED DESCRIPTION:
The goal of this observational study is to investigate the long-term effects of a combined slow and rapid weight reduction strategy on the physiological performance, mental state, and sleep quality of male freestyle wrestlers over the period leading up to a competition. The main question it aims to answer is:

Does the combined weight reduction approach affect the physiological performance, mental state, and sleep quality of male freestyle wrestlers when implemented during the pre-competition phase?

Participants, who are already undergoing this weight reduction strategy as part of their regular training regimen for the 2024 Chinese Wrestling Championships, will be assessed at three distinct time points over a 38-day period. The study will involve the following detailed procedures:

Participant Selection: The study includes 16 male freestyle wrestlers from Sichuan Province, China, with an average age of 20.2 years, and extensive competitive experience.

Study Duration: The observation period spans 38 days prior to the competition, divided into a 30-day slow weight reduction phase and a 7-day rapid weight reduction phase, with the final assessment conducted the day before the competition.

Data Collection: Participants will undergo a series of tests at three time points (T1, T2, T3):

T1: First day of slow weight reduction. T2: First day of rapid weight reduction. T3: The day before the competition.

Testing Indicators:

Physiological performance will be measured through heart rate, blood pressure, blood tests for markers like creatine kinase, testosterone, and immunoglobulin G, body composition analysis, and anaerobic power testing.

Mental state will be evaluated using the Profile of Mood States questionnaire, assessing mood dimensions such as tension, anger, fatigue, depression, energy, confusion, and self-esteem.

Sleep quality will be assessed using the Pittsburgh Sleep Quality Index, a questionnaire that evaluates sleep quality over the past month.

Data Analysis: The study will analyze changes in physiological performance, mental state, and sleep quality from T1 to T3, looking for significant differences that may indicate the impact of the weight reduction strategy.

Ethical Considerations: The study is approved by the Ethics Committee for Human Experiments at Sichuan Sports College and adheres to the Declaration of Helsinki. All participants provide informed consent.

Study Hypothesis: There will be significant differences in the changes in physiological performance, mental state, and sleep quality of male freestyle wrestlers during the pre-competition slow and rapid weight reduction training period.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be male freestyle wrestlers aged 18 years or older
* Athletes should be preparing for the 2024 Chinese Wrestling Championships
* Individuals must be willing to undergo all tests and assessments at the three specified time points (T1, T2, T3) over the 38-day study period
* Participants should be in good health, with no medical conditions that would prevent them from completing the study
* Athletes must be undergoing a combined slow and rapid weight reduction strategy as part of their regular training regimen

Exclusion Criteria:

* Individuals with a history of severe cardiovascular, metabolic, or endocrine disorders that could affect the study outcomes
* Wrestlers who are unable to comply with the study's testing schedule or intervention protocols
* Participants with any condition that would make them unsuitable for the anaerobic power testing or blood sampling
* Wrestlers who are unwilling or unable to provide informed consent

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2024-03-26 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-05-03 (Actual)

PRIMARY OUTCOMES:
Blood Pressure Testing | 38 days
  Participants' blood pressure were measured in a supine position using an instrument (manufactured in Shenzhen, China, model: CK-W355) by laboratory personnel, with the average of three readings taken.
Serum testosterone | 38 days
  Approximately 3 mL of antecubital venous blood was collected from participants and tested for serum testosterone.
Serum creatine kinase | 38 days
  Approximately 3 mL of antecubital venous blood was collected from participants and tested for serum creatine kinase.
Serum blood urea | 38 days
  Approximately 3 mL of antecubital venous blood was collected from participants and tested for serum blood urea.
Serum immunoglobulin G | 38 days
  Approximately 3 mL of antecubital venous blood was collected from participants and tested for serum immunoglobulin G.
Serum immunoglobulin A | 38 days
  Approximately 3 mL of antecubital venous blood was collected from participants and tested for serum immunoglobulin A.
Serum immunoglobulin M | 38 days
  Approximately 3 mL of antecubital venous blood was collected from participants and tested for serum immunoglobulin M.
Body Composition Testing | 38 days
  The participants' weight and body fat percentage were tested using the Korean INBODY 3.0.
The Profile of Mood States | 38 days
  For psychological state: the Profile of Mood States, a tool for studying mood states and their relation to exercise performance, was used. Participants answered 40 questions with a five-point scale (0 to 4 points, with 0 indicating 'almost none', 1 'a little', 2 'moderate', 3 'quite a bit', and 4 'extremely'), including seven mood dimensions: tension, anger, fatigue, depression, energy, confusion, and self-esteem. Energy and self-esteem are positive mood dimensions, with higher scores indicating better mood states, while the other five are negative mood dimensions, with higher scores indicating worse mood states. The total score, total mood disturbance (calculated as the sum of the five negative mood scores minus the sum of the two positive mood scores plus 100), indicates worse mood states with higher scores. The scale has a reliability between 0.60 and 0.82 and a validity greater than 0.90 for Chinese individuals.
Sleep quality | 38 days
  The pittsburgh sleep quality index, a questionnaire for assessing sleep quality over the past month, consists of 18 self-rated items forming seven components, with a total score ranging from 0 to 21, where higher scores indicate worse sleep quality. The scale has a reliability between 0.65 and 0.84 and a validity greater than 0.85 for Chinese individuals.
Anaerobic Power Testing | 38 days
  The Wingate 30-second anaerobic test (MONARK 894E, MONARK Company, Sweden) was used. Participants pedalled as fast as possible, adjusting to the prescribed resistance load within 3 to 4 seconds, and started timing for a 30-second all-out cycling exercise. The average power over 30 seconds, total work output, maximum power output within 5 seconds, and minimum power output within 5 seconds were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Xiong Weizhi, Dr, Study Chair — Chengdu Sport University
Locations (1):
- Chengdu Sport University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No